CLINICAL TRIAL: NCT05297643
Title: Effects of Extracorporeal Shock Wave Therapyy Added To Complex DecongestiveTherapy In Patient With Breast Cancer Releated Lymphedema
Brief Title: Effects of Extracorporeal Shock Wave Therapy Added To Complex DecongestiveTherapy In Patıent With Lymphedeme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Assistant professor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Lymphedema, Breast Cancer
Keywords: Lymphedema; Complex DecongestiveTherapy; Extracorporeal Shock Wave Therapy
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema

STUDY DESIGN:
Intervention Model Description: randomized controlled trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A Complex decongestive treatment program consisting of manual lymphatic drainage, compression therapy, skin care and remedal exercise will be applied to the patients in this group. Exercise progame includes breathing exercises, joint range of motion exercise, pumping, stretching exercises and aerobic exercises( same with control grup).
  In addition, ESWT will be applied as 2 sessions in the first two weeks and 1 session in the 3rd week. In ESWT, 2500 shocks will be applied per session with a frequency of 4 Hz at 2 bar pressure while the patient is in the supine position.
  The distribution of this treatment is planned to be 750 shocks to the axillary lymph nodes and 250 shocks to the cubital lymph nodes.
  The remaining 1500 shocks will be applied to the arm, forearm, and hand. While determining the dose and duration of ESWT to be applied in the study, it was arranged to be similar to the studies and reviews in the literature.
  Interventions: Device: Ekstracorporeal Shock Wave Therapy (ESWT); Other: complex decongestive therapy
- control group (Other): A Complex decongestive treatment program consisting of manual lymphatic drainage, compression therapy, skin care and remedal exercise will be applied to the patients in this group. Exercise progame includes breathing exercises, joint range of motion exercise, pumping, stretching exercises and aerobic exercises
  Interventions: Other: complex decongestive therapy

INTERVENTIONS:
Device: Ekstracorporeal Shock Wave Therapy (ESWT) — Extracorporeal Shock Wave Therapy (ESWT); It is a treatment method in which high-intensity pressure waves are applied to the desired point in the body. It has been used in the treatment of kidney stones in previous years, and changes in bone tissue have been observed (12). Today, it is used in musculoskeletal system diseases such as plantar fasciitis, epicondylitis, achiltendinitis, osteoarthritis
  Arms: Experimental Group
Other: complex decongestive therapy — Complex decongestive therapy consists of manual lymphatic degeneration, compression therapy, skin care and remedal exercise.

SUMMARY:
Extracorporeal Shock Wave Therapy (ESWT); It is a treatment method in which high-intensity pressure waves are applied to the desired point in the body. It has been used in the treatment of kidney stones in previous years, and changes in bone tissue have been observed . Today, it is used in musculoskeletal diseases such as plantar fasciitis, epicondylitis, achillestendinitis, and osteoarthritis. The main mechanism of action of ESWT is not clearly known, but many studies have shown that it stimulates the early release of angiogenesis-related growth factors such as endothelial nitric oxide synthase (eNOS) and vascular endothelial growth factor (VEGF) and increases blood circulation with induced neovascularization, resulting in cell proliferation and tissue growth. It has been shown to increase regeneration . It has been found to be effective in lymphedema with neovascularization and lymphatic channel synthesis . In the literature, there are studies investigating the additional contributions of complex decongestive therapy combined with ESWT in patients with lymphedema.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women and the leading cause of death in the world. With the advances in early diagnosis and treatment methods, the mortality rate in breast cancer tends to decrease . However, some complications secondary to both the disease and the treatment can be seen in patients who have received treatment. Examples of these complications are; functional disability, advanced peripheral neuropathy secondary to chemotherapy agents, pain, weight loss or weight gain, depression, lymphedema. lymphedema; It is primarily a condition characterized by abnormal accumulation of fluid in the subcutaneous tissue and subfascial layer. Lymphedema occurs as a result of fluid accumulation above the lymphatic carrying capacity or insufficient lymphatic transport. Lymphedema is a chronic progressive disease. Therefore, early diagnosis and treatment are important to prevent complications (disability, infection, depression, pain, malignant transformation).

Lymphedema secondary to breast cancer was first defined as postmastectomy lymphedema by Hastead in 1921. Treatment of secondary lymphedema is multidisciplinary. The gold standard method is complex decongestive therapy (CDT). It consists of two phases. Phase 1: lasting 2-6 weeks; manual lymphatic drainage (MLD), multilayer bandaging, exercise and skin care. With MLD treatment, fluid is removed and bandaging is applied to prevent re-accumulation. Exercise and skin care are explained to the patient. When the plateau phase is reached in the measurements, the protection phase is started. Phase 2: includes self-massage, exercise, skin care, bandaging and the use of compression garments. Apart from these; Low-dose laser, oral medications, pneumatic compression devices and surgical methods can be used in the treatment of lymphedema. In this study, both groups will receive MLD treatment. In other words, no group will be left without treatment.

Extracorporeal Shock Wave Therapy (ESWT); It is a treatment method in which high-intensity pressure waves are applied to the desired point in the body. It has been used in the treatment of kidney stones in previous years, and changes in bone tissue have been observed. Today, it is used in musculoskeletal diseases such as plantar fasciitis, epicondylitiS and osteoarthritis. The main mechanism of action of ESWT is not clearly known, but many studies have shown that it stimulates the early release of angiogenesis-related growth factors such as endothelial nitric oxide synthase (eNOS) and vascular endothelial growth factor (VEGF) and increases blood circulation with induced neovascularization, resulting in cell proliferation and tissue growth. It has been shown to increase regeneration . It has been found to be effective in lymphedema with neovascularization and lymphatic channel synthesis . In the literature, there are studies investigating the additional contributions of complex decongestive therapy combined with ESWT in patients with lymphedema. While planning this study, the dose and duration of ESWT were determined based on these studies.

ELIGIBILITY:
Inclusion Criteria:

1. Be over 18 years old
2. History of lymphedema for at least 6 months after breast cancer treatment
3. Ending radiotherapy treatment at least 2 months ago
4. Not being included in the Complex DecongestiveTherapy program within 3 months
5. Having unilateral lymphedema
6. Having stage 2 lymphedema
7. Signing of the voluntary consent form
8. Patients who have undergone oncological follow-up for breast cancer in the last 6 months and have been shown to be free of recurrence and metastasis

Exclusion Criteria:

1. Active cancer
2. Skin infection, radiotherapy burn
3. Severely affected upper extremity range of motion 4 kidney failure

5. Heart failure 6. History of untreated deep venous thrombosis 7. Body mass index I≥35 kg/m2 8. Using a pacemaker/internal defibrillator 9. Patients continuing radiotherapy and/or chemotherapy treatment 10. Having bilateral lymphedema 11. Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — BREAST CANCER-RELATED LYMPHEDEMA ONLY OCCUR IN WOMEN
Enrollment: 44 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Pain; | Baseline
  Evaluation of Pain;
  Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Evaluation of Pain; | 3th week (after treatment)
  Evaluation of Pain;
  Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Evaluation of Pain; | 12th week
  Evaluation of Pain;
  Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Environmental Measurement; | Baseline
  Both upper extremities of the patient will be measured with the help of a tape measure. The cm difference between both upper extremities will be recorded. Measurements will be made from the MCP (metacarpophalangeal joint), wrist, lateral epicondyle, and 10 cm above and below the lateral epicondyle.
Environmental Measurement; | 3th week (after treatment)
  Both upper extremities of the patient will be measured with the help of a tape measure. The cm difference between both upper extremities will be recorded. Measurements will be made from the MCP (metacarpophalangeal joint), wrist, lateral epicondyle, and 10 cm above and below the lateral epicondyle.
Environmental Measurement; | 12th week
  Both upper extremities of the patient will be measured with the help of a tape measure. The cm difference between both upper extremities will be recorded. Measurements will be made from the MCP (metacarpophalangeal joint), wrist, lateral epicondyle, and 10 cm above and below the lateral epicondyle.

SECONDARY OUTCOMES:
Shoulder and Hand Questionnaire (Quick-DASH) | Baseline
  The short version of the Arm, Shoulder and Hand Questionnaire (Quick-DASH) Disability will be used to evaluate the functional status of the patients. Quick-DASH is a self-report questionnaire designed to measure physical function and symptoms in people with upper extremity musculoskeletal conditions.
Shoulder and Hand Questionnaire (Quick-DASH) | 3th week (after treatment)
  The short version of the Arm, Shoulder and Hand Questionnaire (Quick-DASH) Disability will be used to evaluate the functional status of the patients. Quick-DASH is a self-report questionnaire designed to measure physical function and symptoms in people with upper extremity musculoskeletal conditions.
Shoulder and Hand Questionnaire (Quick-DASH) | 12th week
  The short version of the Arm, Shoulder and Hand Questionnaire (Quick-DASH) Disability will be used to evaluate the functional status of the patients. Quick-DASH is a self-report questionnaire designed to measure physical function and symptoms in people with upper extremity musculoskeletal conditions.
Measurement of Joint Range of Motion: | Baseline
  Measurement of shoulder joint range of motion (ROM) with goniometer is the most frequently used method that provides objective evaluation and error-free measurement in clinical practice. In our study, shoulder ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Measurement of Joint Range of Motion: | 3th week (after treatment)
  Measurement of shoulder joint range of motion (ROM) with goniometer is the most frequently used method that provides objective evaluation and error-free measurement in clinical practice. In our study, shoulder ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Measurement of Joint Range of Motion: | 12th week
  Measurement of shoulder joint range of motion (ROM) with goniometer is the most frequently used method that provides objective evaluation and error-free measurement in clinical practice. In our study, shoulder ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Grip Strength: | Baseline
  Goarse grip; It is caused by the combined activities of the intrinsic and extrinsic muscles of the hand. In our study, Jamar dynamometer was used for the evaluation of rough grip strength. The digital handheld dynamometer can measure in pounds and kg.
Grip Strength: | 3th week (after treatment)
  Goarse grip; It is caused by the combined activities of the intrinsic and extrinsic muscles of the hand. In our study, Jamar dynamometer was used for the evaluation of rough grip strength. The digital handheld dynamometer can measure in pounds and kg. .
Grip Strength: | 12th week
  Goarse grip; It is caused by the combined activities of the intrinsic and extrinsic muscles of the hand. In our study, Jamar dynamometer was used for the evaluation of rough grip strength. The digital handheld dynamometer can measure in pounds and kg.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Asst Prof, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University Faculty of Medicine, Kırşehir, City Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cebicci MA, Sutbeyaz ST, Goksu SS, Hocaoglu S, Oguz A, Atilabey A. Extracorporeal Shock Wave Therapy for Breast Cancer-Related Lymphedema: A Pilot Study. Arch Phys Med Rehabil. 2016 Sep;97(9):1520-1525. doi: 10.1016/j.apmr.2016.02.019. Epub 2016 Mar 15. PMID 26987620
- [Result] Lee KW, Kim SB, Lee JH, Kim YS. Effects of Extracorporeal Shockwave Therapy on Improvements in Lymphedema, Quality of Life, and Fibrous Tissue in Breast Cancer-Related Lymphedema. Ann Rehabil Med. 2020 Oct;44(5):386-392. doi: 10.5535/arm.19213. Epub 2020 Sep 28. PMID 32986941
- [Result] Joos E, Vultureanu I, Nonneman T, Adriaenssens N, Hamdi M, Zeltzer A. Low-Energy Extracorporeal Shockwave Therapy as a Therapeutic Option for Patients with a Secondary Late-Stage Fibro-Lymphedema After Breast Cancer Therapy: A Pilot Study. Lymphat Res Biol. 2021 Apr;19(2):175-180. doi: 10.1089/lrb.2020.0033. Epub 2020 Aug 11. PMID 32780632
- [Result] Bae H, Kim HJ. Clinical outcomes of extracorporeal shock wave therapy in patients with secondary lymphedema: a pilot study. Ann Rehabil Med. 2013 Apr;37(2):229-34. doi: 10.5535/arm.2013.37.2.229. Epub 2013 Apr 30. PMID 23705118